### ATH-1017-AD-0203 OLEX Analysis Summary

| Sponsor: | Athira Pharma, Inc. |
|---|---|
| Sponsor Address: | 18706 North Creek Parkway<br>Suite 104<br>Bothell, WA 98011 |
| Protocol Number: | ATH-1017-AD-0203 Open Label Extension Study |
| Study Title | Open-Label Extension of Studies ATH-1017-AD-0201 and ATH-1017-AD-0202 in Subjects with Mild to Moderate Alzheimer's Disease |
| <b>Document Version:</b> | V1.1 |
| Version Date: | December 05, 2024 |

## **Confidentiality Statement**

This document contains confidential and proprietary information, and is not to be distributed to any third party

### **Approvals**

| Signature/Date: |
|-----------------|

| Reviewed By: | Signature/Date: |
|--------------|-----------------|

Document History - Changes Compared to Previous Version

| Version | Date | Changes |
|---|---|---|
| 1.0 | 02Oct2024 | Initial Version |
| | | Added 4 Listings, 1 Figure and updated footnotes for some outputs to note participants might be counted for both dose |
| 1.1 | 05Dec2024 | groups. |

ATH-1017-AD-0203 OLEX Analysis Summary Athira Pharma, Inc. ATH-1017 Program Version 1.1

## **TABLE OF CONTENTS**

| TABLE OF CONTENTS | 4 |
|-----------------------------------|---|
| ABBREVIATIONS | 5 |
| 1 INTRODUCTION AND SCOPE | 6 |
| 2 TLF TABLE OF CONTENTS | 6 |
| 3 TLF DRY RUN APPROACH | 7 |
| ATTACHMENT A – TLF SPECIFICATIONS | 8 |

### **ABBREVIATIONS**

| AE | Adverse Event |
|-------|-----------------------------------------------|
| AD | Alzheimer's Disease |
| ApoE | Apolipoprotein E |
| ERP | Event related potential |
| FDA | Food and Drug Administration |
| FPI | First Patient In |
| FTP | File Transfer Protocol |
| GCP | Good Clinical Practice |
| MMSE | Mini-Mental State Examination |
| QC | Quality Control |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SPO | Share Point Online |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TMF | Trial Master File |
| TLFs | Tables, Listings, and Figures |

### 1 INTRODUCTION AND SCOPE

The purpose of this Analysis Summary is to describe the framework for the reporting, summarization and statistical analysis methodology of the safety parameters measured throughout the study.

As the study was terminated by the Sponsor, only a basic set of safety tables, listings and figures will be generated.

As per the protocol, the baseline flag will be assigned to the Visit 8 assessment from parent study for the participants who entered in OLEX without the time gap and then to the Rollover Visit 2 Day 1 assessment from the OLEX study for the subject who entered in OLEX with Gap >= 30 days.

If Visit 8 and Visit 9 records are missing in the parent study for a participant, the baseline value will be considered missing. Therefore, those specific participants will be excluded from change from baseline calculations.

Due to strict database lock timelines, any minor updates to TLF shells post-signature will not require a new version of this Analysis Plan.

### 2 TLF TABLE OF CONTENTS

| | AD-203 OLEX |
|---|---|
| Output Title Type/Number | |
| Table 14.1.1.4 | Participant Disposition, Early Withdrawal from the Study |
| Table 14.1.1.5 | Major Protocol Deviations |
| Table 14.1.2.1 | Demographics and Baseline Characteristics |
| Table 14.1.4.1 | Duration of Exposure to Study Treatment |
| Table 14.3.1.1 | Overall Summary of Adverse Events |
| Table 14.3.1.2 | Treatment Emergent Adverse Events by Primary System Organ Class and Preferred Term |
| Table 14.3.1.3 | Treatment-Related TEAEs by Primary System Organ Class and Preferred Term |
| Table 14.3.1.4 | Serious TEAEs by Primary System Organ Class and Preferred Term |
| Table 14.3.1.5 | Treatment-Related Serious TEAEs by Primary System Organ Class and Preferred Term |
| Table 14.3.1.6 | Adverse Events Leading to Study Drug Withdrawal by Primary System Organ Class and Preferred Term |
| Table 14.3.1.7 | Adverse Events Leading to Study Drug Interruption by Primary System Organ Class and Preferred Term |
| Table 14.3.1.8 | Treatment Emergent Adverse Events by Primary System Organ Class, Preferred Term, and Maximum Severity |
| Table 14.3.1.9 | Injection Site Reactions by Preferred Term |
| Table 14.3.4.3 | Hematology Shift from Baseline to Worst Post-Baseline Values |
| Table 14.3.4.6 | Chemistry Shift from Baseline to Worst Post-Baseline Values |

| AD-203 OLEX | |
|---|---|
| Output<br>Type/Number | Title |
| Table 14.3.4.9A | Urinalysis Shift from Baseline to Worst Post-Baseline Values (Normal/Abnormal) |
| Table 14.3.4.9B | Urinalysis Shift from Baseline to Worst Post-Baseline Values (Low/Normal/High) |
| Table 14.3.7.9 | Summary of Liver Related Laboratory Abnormalities |
| Table 14.3.7.11 | Summary of Eosinophil Lab Abnormalities |
| Table 14.3.6.2 | Potential Vital Signs Values of Concern at Any Time Post-Baseline |
| Table 14.3.7.4 | ECG Interpretation at Any Time Post-Baseline |
| Table 14.3.7.5 | Shifts from Baseline to Post-Baseline in ECG Values |
| Table 14.3.7.6 | Potential ECG Values of Concern at Any Time Post-Baseline |
| Table 14.3.8.2 | Concomitant Medications by ATC Class and Preferred Name |
| Listing 14.3.2.1 | Deaths Reported |
| Listing 14.3.2.2 | Serious Adverse Events |
| Listing 14.3.2.3 | Adverse Events |
| Listing 16.2.1 | Participant Disposition |
| Listing 16.2.1.1 | Participants Reduced to 40mg Dose |
| Listing 16.2.2 | Major Protocol Deviations |
| Listing 16.2.4.1 | Participant Demographics and Baseline Characteristics |
| Listing 16.2.6 | Prior and Concomitant Medications |
| Listing 16.2.8.1 | Chemistry Laboratory Values Where at Least One Value is a Potential Value of Concern |
| Listing 16.2.8.2 | Hematology Laboratory Values Where at Least One Value is a Potential Value of Concern |
| Listing 16.2.8.3 | Vital Signs Values Where at Least One Value is a Potential Value of Concern |
| Listing 16.2.9 | ECG Parameters Where at Least One Value is a Potential Value of Concern |
| Figure 14.3.1.1 | eDISH (evaluation of Drug Induced Serious Hepatotoxicity) |

### 3 TLF DRY RUN APPROACH

No formal Dry Run is or will be scheduled prior to database lock. Once database lock occurs, the TLFs specified in the Table of Contents and Attachment A will be refreshed. MMS will internally review the TLFs prior to delivery to Athira. Once the TLFs and datasets are delivered to Athira, they will be considered Post-DBL Draft 1. Athira will have an opportunity to comment and make slight adjustments via the comment log on the SharePoint site. A Comment Resolution Meeting (CRM) will be scheduled between the main points of contact from both parties, if needed. MMS will consider all comments and will update the TLFs accordingly. Changes to the approved TLF specifications, requests for additional/new outputs, and/or programmatic updates to resolve data issues will incur additional cost and may impact the timeline. The next delivery of TLFs / datasets will be considered Final.

### ATTACHMENT A – TLF SPECIFICATIONS

### ICH E3 TLG NUMBERING GUIDELINE

• Guideline for Industry: Structure and Content of Clinical Study Reports

This is a summary of the guideline as it applies to numbering tables, listings and graphs for programmers and statisticians. To ensure most current guideline is being followed, reference the link on fda.gov. https://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformation/guidances/ucm073113.pdf

- Section 14.x TABLES, FIGURES, AND GRAPHS REFERRED TO BUT NOT INCLUDED IN THE TEXT
  - o 14.1 Demographic Data Summary figures and tables
  - o 14.2 Efficacy Data Summary figures and tables
  - o 14.3 Safety Data Summary figures and tables
  - o 14.3.1 Displays of Adverse Events
  - o 14.3.2 Listings of Deaths, Other Serious and Significant Adverse Events
  - o 14.3.3 Narratives of Deaths, Other Serious and Certain Other Significant Adverse Events
  - o 14.3.4 Abnormal Laboratory Value Listing (each patient)
- Section 16.x APPENDICES
  - o 16.1 Study Information
  - o 16.2 Patient Data Listings
    - 16.2.1 Discontinued participants
    - 16.2.2 Protocol deviations
    - 16.2.3 Participants excluded from the efficacy analysis
    - 16.2.4 Demographic data
    - 16.2.5 Compliance and/or drug concentration data (if available)
    - 16.2.6 Individual efficacy response data
    - 16.2.7 Adverse event listings (each patient)
    - 16.2.8 Listing of individual laboratory measurements by patient, when required by regulatory authorities
  - o 16.3. Case Report Forms (CRF's)
    - 16.3.1 CRF's for deaths, other serious adverse events, and withdrawals for adverse events
    - 16.3.2 Other CRF's submitted
  - o 16.4 Individual Patient Data Listings
- If there are multiple listings that belong in one of the ICH appendix sections, the number format should be 16.2.X.Y. (X=ICH number listed above, Y = sequential number). Example, if there are 5 AE listings then they would be number 16.2.7.1 to 16.2.7.5. If there is only one, then use 16.2.7.

# DISPOSITION, DEMOGRAPHICS, AND BASELINE CHARACTERISTICS

# Table 14.1.1.4 Participant Disposition, Early Withdrawal from the Study Safety Population

| Disposition/<br>Reason | 40 mg ATH-1017<br>n (%) | 70 mg ATH-1017<br>n (%) | Overall<br>n (%) |
|---|---|---|---|
| Safety population | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ongoing Study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed Study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued Study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary reason for discontinuation of the study - n (%) | | | |
| Any Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lack of Efficacy | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal by Subject or Legally Authorized Representative (LAR) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Physician Decision | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Non-Compliance with Study Drug | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Site Terminated by Sponsor | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Repeat incapacity of subject and/or caregiver (in the judgement of the investigator to properly administer drug) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Prolonged or definitive loss of caregiver without adequate seplacement | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Nursing home replacement | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to Follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week of Early Withdrawal | | | |
| 0-2 Weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2-4 Weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 32-34 Weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MISSING END OF STUDY DATE | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- Percentages are calculated using the number of participants in each treatment group as the denominator.
- Participants receiving both 40 mg and 70 mg are counted in both dose groups; Overall is not a summation of the dose groups.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y

NOTE: Ensure that the primary reason for discontinuation of study listed in the shell matches the options in the CRF.

### Programming Notes:

• Week of Early Withdrawal displayed in the interval of 2 weeks till last available week data.


# Table 14.1.1.5 Major Protocol Deviations Safety Population

| Major Protocol Deviation/ Reasons | 40 mg ATH-1017<br>(N=xxx)<br>n(%) | 70 mg ATH-1017<br>(N=xxx)<br>n(%) | Overall (N=xxx) n(%) |
|---|---|---|---|
| Number of participants with at least 1 major protocol deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Inclusion/Exclusion Criteria | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Informed Consent Procedures | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Study Procedures | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit Schedule/Interval | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> A participant with multiple protocol deviations within a deviation category or deviation term is counted only once.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y

Version: DRAFT

#### Programming Notes:

• Please add all the possible major protocol reasons as per the data collected.

<sup>-</sup> Participants may have multiple protocol deviations.

<sup>-</sup> Participants with a reported major protocol deviation in 70mg will be counted in the 70mg column. If that same participant switched to 40mg and reported a major protocol deviation during the 40mg timeframe, that new major protocol deviation is reported in the 40mg column. If the same major protocol deviation reported while taking 40mg and 70mg then it is counted in both 40mg and 70mg groups; Overall is not a summation of the dose groups.

<sup>-</sup> If deviation start date is missing, the deviation is counted in each dose groups.

Table 14.1.2.1
Demographics and Baseline Characteristics
Safety Population

| Parameter | 40 mg ATH-1017 | 70 mg ATH-1017 | Overall |
|---|---|---|---|
| Statistic | (N=xxx) | (N=xxx) | (N=xxx) |
| Age at Informed Consent (years) | | | |
| n | XXX | xxx | XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | xx.x | XX.X |
| (Q1, Q3) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Min, Max | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X |
| P-value | x . x | XXX | |
| Age Group - n(%) | | | |
| <65 years | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 65 years | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Available | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| P-value | X.X | XXX | |
| Ethnicity - n(%) | | | |
| Hispanic Or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic Or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Specified | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Available | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| P-value | X.X | XXX | |
| Race - n(%) | | | |
| American or Alaskan Native | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Black | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hawaiian or Pacific Islander | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| White | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Available | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| American or Alaskan Native | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| P-value | X • X | XXX | |
| Sex - n(%) | | | |
| Male | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Available | | | |
| P-value | X • X | xxx | |

| Parameter Statistic | 40 mg ATH-1017<br>(N=xxx) | 70 mg ATH-1017<br>(N=xxx) | Overall<br>(N=xxx) |
|---|---|---|---|
| | (IV AAA) | (IV AAA) | (II AAA) |
| Years of Education | | | |
| n | XXX | xxx | XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | xx.x | XX.X |
| (Q1, Q3) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Min, Max | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X |
| P-value | X • X | XXX | |
| Height (cm) | | | |
| n | XXX | xxx | XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X |
| (Q1, Q3) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Min, Max | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |
| P-value | х.х | XXX | |
| Weight (kg) | | | |
| n | XXX | XXX | XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | XX.X | XX.X |
| (Q1, Q3) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Min, Max | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |
| P-value | X • X | x.xxxx | |
| Body Mass Index (kg/m²) | | | |
| n | XXX | xxx | XXX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | xx.x | XX.X |
| (Q1, Q3) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| P-value | x.x | | · |

<sup>-</sup> SD: Standard Deviation, Q1: 1st Quartile, Q3: 3rd Quartile; n: number of participants with values for given treatment group.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

<sup>-</sup> Percentages are calculated using the number of participants in each treatment group as the denominator.

<sup>-</sup> MMSE Severity = Mild if MMSE total Score is between 20-24. MMSE Severity = Moderate if MMSE total Score is between 14-19.

<sup>-</sup> p-values presented test for a difference between participants who received 40mg ATH-1017 and participants who received 40mg ATH-1017. A 2 sample t-test is used to test the difference for continuous variables and a chi-squared test of independence is used to test the difference for categorical variables. N: number of Participants in the specified population without Acetylcholinesterase Inhibitors for given treatment group. Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.

# Exposure

Table 14.1.4.1
Duration of Exposure to Study Treatment
Safety Population

| Category | 40 mg ATH-1017<br>(N=xxx) | 70 mg ATH-1017<br>(N=xxx) | Overall<br>(N=xxx) |
|---|---|---|---|
| Duration of study treatment (days) | | | |
| n | | | |
| Mean | XX | XX | XX |
| SD | XX.X | XX.X | XX.X |
| Min | XX.XX | XX.XX | xx.xx |
| Median | XX | xx | XX |
| Q1,Q3 | XX.X | xx.x | xx.x |
| Max | xx,xx | xx,xx | xx,xx |
| | XX | xx | xx |
| Duration of exposure, n(%) At least 1 dose | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 days to <4 weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 weeks to <8 weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 8 weeks to <12 weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 12 weeks to <16 weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 16 weeks to <20 weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 20 weeks to <24 weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 24 weeks to <48 weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 48 weeks to <72 weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 72 weeks to <96 weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 96 weeks or more | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- SD: Standard Deviation, Q1: 1st Quartile, Q3: 3rd Quartile
- Day is relative to first dose date.
- Duration of Exposure (Days) defined as date of last dose date of first dose +1
- Participants receiving both 40 mg and 70 mg are counted in both dose groups for their respective time in each dose group; Overall is not a summation of the dose groups.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y

### Programming Notes:

• Duration of Exposure (Days) defined as date of last dose - date of first dose +1. For participants ongoing at time of the data cut, the date of cut-off was used as the date of last dose.

## **SAFETY DATA**

**Displays of Adverse Events** 


# Table 14.3.1.1 Overall Summary of Adverse Events Safety Population

| | 40 mg ATH-1017<br>(N=xxx)<br>n(%) | 70 mg ATH-1017<br>(N=xxx)<br>n(%) | Overall<br>(N=xxx)<br>n(%) |
|---|---|---|---|
| Number of participants with at least 1 AE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of participants with at least 1 TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of participants with at least 1 Treatment-Related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Participants with serious or other significant TEAEs | | | |
| Death SAE(s) Treatment-Related Serious TEAE(s) TEAEs Leading to Study Drug Withdrawal TEAEs Leading to Study Drug Interruption | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

<sup>-</sup> AE: Adverse Event; TEAE: Treatment Emergent Adverse Event; SAE: Serious Adverse Event. N: number of Participants in the specified population for given treatment group. Related includes related, probably related, and possibly related events.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


Programming Notes:

•

<sup>-</sup> Percentages are based on the Safety Population; Deaths are AEs with reported outcome of Fatal.

<sup>-</sup> All AE terms were coded to Medical Dictionary for Regulatory Activities Terminology (MedDRA®) version 24.0.

<sup>-</sup> Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.

<sup>-</sup> Participants with a reported AE in 70mg will be counted in the 70mg column. If that same participant switched to 40mg and reported an AE during the 40mg timeframe, that new AE is reported in the 40mg column. If the same event reported while taking 40mg and 70mg then it is counted in both 40mg and 70mg groups; Overall is not a summation of the dose groups.


 ${\tt Table~14.3.1.2}$  Treatment Emergent Adverse Events by Primary System Organ Class and Preferred Term Safety Population

| System Organ Class (SOC)<br>Preferred Term (PT) | 40 mg ATH-1017<br>(N=xxx)<br>n (%) | 70 mg ATH-1017<br>(N=xxx)<br>n (%) | Overall<br>(N=xxx)<br>n (%) |
|---|---|---|---|
| Number of participants with at least 1 TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- TEAE: Treatment Emergent Adverse Event; n = number of participants with at least one TEAE occurring; % = (n/N) \*100; N: number of participants in the specified population for given treatment group. Percentages based on Safety Population. SOCs are presented alphabetically; PTs are sorted by decreasing frequency in the Overall column. A participant with multiple adverse events within a primary SOC and PT is counted only once for raw incidence rates. All AE terms were coded to Medical Dictionary for Regulatory Activities Terminology (MedDRA®) version 24.0. Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received. Participants with a reported AE in 70mg will be counted in the 70mg column. If that same participant switched to 40mg and reported an AE during the 40mg timeframe, that new AE is reported in the 40mg column. If the same event reported while taking 40mg and 70mg then it is counted in both 40mg and 70mg groups; Overall is not a summation of the dose groups.

Generated from program.sas on DDMMMYYYY HH:MM Data as of: DDMMYYYY

Page X of Y


•

### 

Repeat Table 14.3.1.2 for Treatment-Related TEAEs. Replace first row with "Number of participants with at least 1 Treatment-Related TEAE"

Programming Notes: Add below footnote additionally

- Related includes related, probably related, and possibly related events.

#### 

Use the Table 14.3.1.2 shell.

Replace first row with "Number of participants with at least 1 Serious TEAE" NOTE: subset this table to show Serious TEAEs.

Programming Notes:

Table 14.3.1.5

Treatment-Related Serious TEAEs by Primary System Organ Class and Preferred Term Safety Population

Use the Table 14.3.1.2 shell.

Replace first row with "Number of participants with at least 1 Treatment-Related Serious TEAE" NOTE: subset this table to show Treatment-Related Serious TEAEs.

Programming Notes: Add below footnote additionally

- Related includes related, probably related, and possibly related events.

Table 14.3.1.6

Adverse Events Leading to Study Drug Withdrawal by Primary System Organ Class and Preferred Term Safety Population

Use the Table 14.3.1.2 shell.

Replace first row with "Number of participants with at least 1 AE leading to study drug withdrawal" NOTE: subset this table to show AEs leading to study drug discontinuation only.

Programming Notes:

•

 ${\tt Table~14.3.1.7}$  Adverse Events Leading to Study Drug Interruption by Primary System Organ Class and Preferred Term Safety Population

Use the Table 14.3.1.2 shell. Replace first row with "Number of participants with at least 1 AE leading to study drug interruption"

NOTE: subset this table to show AEs leading to study drug interruption only.

Programming Notes:

•

Athira Pharma, Inc.

ATH-1017-AD-0203


| Primary System Organ Class (SOC)/<br>Preferred Term (PT) | Severity | 40 mg ATH-1017<br>(N=xxx)<br>n(%) | 70 mg ATH-1017<br>(N=xxx)<br>n(%) | Overall (N=xxx) n(%) |
|---|---|---|---|---|
| Number of participants with at least 1 TEAE | Overall | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System organ class 1 | Overall | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | Overall | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | Overall | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> TEAE: Treatment Emergent Adverse Event. A participant with multiple adverse events within a SOC or PT and a given severity is counted only once n = number of participants with at least one TEAE occurring; % = (n/N) \*100. N: number of participants in the specified population for given treatment group. Percentages are based on the Safety Population. SOCs are presented alphabetically; PTs are sorted within SOC in descending frequency in the 40mg ATH-1017 column. All AE terms were coded to Medical Dictionary for Regulatory Activities Terminology (MedDRA®) version 24.0. Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received. Participants with a reported AE in 70mg will be counted in the 70mg column. If that same participant switched to 40mg and reported an AE during the 40mg timeframe, that new AE is reported in the 40mg column. If the same event reported while taking 40mg and 70mg then it is counted in both 40mg and 70mg groups; Overall is not a summation of the dose groups.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


| Preferred Term (PT) | 40 mg ATH-1017<br>(N=xxx)<br>n (%) | 70 mg ATH-1017<br>(N=xxx)<br>n (%) | Overall<br>(N=xxx)<br>n (%) |
|---|---|---|---|
| Number of participants with at least 1 ISR TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Table 14.3.1.9
Injection Site Reactions by Preferred Term
Safety Population

- ISR = Injection site reaction; TEAE = treatment-emergent adverse event;
- n = number of participants with at least one TEAE occurring; % = (n/N) \*100;
- N: number of participants in the specified population for given treatment group.
- All AE terms were coded to Medical Dictionary for Regulatory Activities Terminology (MedDRA®) version 24.0.
- Participants with a reported ISR in 70mg will be counted in the 70mg column. If that same participant switched to 40mg and reported an ISR during the 40mg timeframe, that new ISR is reported in the 40mg column. If the same ISR reported while taking 40mg and 70mg then it is counted in both 40mg and 70mg groups; Overall is not a summation of the dose groups.

Generated from program.sas on DDMMMYYYY HH:MM Data as of: DDMMYYYY

Page X of Y


#### Programming Notes:

• Table should be sorted by the descending frequency of the ISR PT in the Overall column.

**Listings of Deaths, Other Serious and Significant Adverse Events** 


Listing 14.3.2.1
Deaths Reported
Safety Population

| Treatment | Participant<br>ID | TEAE | Relationship<br>to IMP | AChEI<br>Usage/Age/Sex/<br>Race | Start Date/Time of Study Treatment (Day) | Last Date/Time<br>of Study<br>Treatment (Day) | Death Date/Time (Day) | Reason for Death/<br>Preferred Term |
|---|---|---|---|---|---|---|---|---|
| XXXXXXXX | xxxxxxx | Y | xxxxx | Y/xx/M/<br>xx | YYYY-MM-DD<br>HH:MM (xx) | YYYY-MM-DD<br>HH:MM (xx) | YYYY-MM-DDT<br>HH:MM (xx) | xxxxxxxx/<br>xxxxxxxx |
| XXXXXXXX | xxxxxxx | N | xxxxx | N/xx/F/<br>xx | YYYY-MM-DD<br>HH:MM (xx) | YYYY-MM-DD<br>HH:MM (xx) | YYYY-MM-DDT<br>HH:MM (xx) | xxxxxxxx/<br>xxxxxxxx |

<sup>-</sup> AChEI: Acetylcholinesterase inhibitor; M: Male; F: Female; IMP: Investigational Medicinal Product;

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


Programming Notes:

•

<sup>-</sup> Day is relative to the date of first drug administration.

<sup>-</sup> Missing dates are based on imputed dates (see SAP Appendix 4 for details).

<sup>-</sup> Race Codes: 1: American Indian or Alaska Native; 2: Asian; 3: Black or African American; 4: Native Hawaiian or Other Pacific Islander; 5: White; 6: Other.

<sup>-</sup> All AE terms were coded to Medical Dictionary for Regulatory Activities Terminology (MedDRA®) version 24.0.

<sup>-</sup> Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.


#### Listing 14.3.2.2 Serious Adverse Events Safety Population

| Treatment | Participant<br>ID | | System Organ<br>Class (SOC)/<br>Preferred Term<br>(PT)/<br>Reported Term | Start Date (Day)/<br>End Date (Day) or<br>Ongoing | TEAE | Severity | Treatment Given for AE/ Relationship to IMP/ Relationship to Study Procedure/ Action Taken/ Outcome |
|---|---|---|---|---|---|---|---|
| xxxxxxxx | XXXXXXX | Y/xx/<br>M/<br>xx | xxxx/<br>xxxx/<br>xxxx | YYYY-MM-DD HH:MM (xx)/<br>YYYY-MM-DD HH:MM(xx) | Υ | MILD | Y/ Related/ Related/ Dose not changed/ Recovered/resolved N/ Unrelated/ Related/ Dose not changed/ Recovered/resolved |
| xxxxxxx | xxxxxxx | N/xx/<br>F/<br>xx | xxxx/<br>xxxx/<br>xxxx | YYYY-MM-DD HH:MM (xx)/<br>YYYY-MM-DD HH:MM (xx) | N | MOD | Treatment Given for AE/ Relationship to IMP/ Relationship to Study Procedure/ Action Taken/ Outcome |

<sup>-</sup> TEAE: Treatment Emergent Adverse Event; IMP: Investigational Medicinal Product; AChEI: Acetylcholinesterase inhibitor; M: Male; F: Female.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


Programming Notes:

.

<sup>-</sup> Race Codes: 1: American Indian or Alaska Native; 2: Asian; 3: Black or African American; 4: Native Hawaiian or Other Pacific Islander; 5: White; 6: Other.

<sup>-</sup> Day is relative to the date of first drug administration.

<sup>-</sup> All AE terms were coded to Medical Dictionary for Regulatory Activities Terminology (MedDRA®) version 24.0.

<sup>-</sup> Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.

Athira Pharma, Inc.

ATH-1017-AD-0203


Listing 14.3.2.3
Adverse Events
Safety Population

Use the Listing 14.3.2.2 shell

Programming Notes: Repeat for AEs

•

### **Laboratory Results**

Consider the following decimal precision as a guide for the mean for each parameter, if reported in SI units.

| Parameter | Decimal Precision for Mean |
|---|---|
| Hematology: Hemoglobin, platelets | 1 |
| Chemistry: sodium, chloride, bicarbonate, creatinine, protein, albumin, ALT, AST, GGT, ALP, CK, LDH | |
| Hematology: erythrocytes, leukocytes, lymphocytes, neutrophils, basophils/leukocytes, | 2 |
| eosinophils/leukocytes, lymphocytes/leukocytes, monocytes/leukocytes, neutrophils/leukocytes | |
| Chemistry: potassium, glucose (fasting and non-fasting), urea nitrogen, total bilirubin (total, direct, | |
| indirect), triglycerides, cholesterol (total, LDL, HDL) | |
| Coagulation: prothrombin time, INR, APTT | |
| Hematology: Hematocrit, basophils, eosinophils, monocytes | 3 |
| Chemistry: calcium, phosphate | |
| Note: | |
| • $SD = mean + 1$ , | |
| • Median = mean | |
| • $Min/Max = mean - 1$ | |

Chemistry results are usually displayed in alphabetical order. For hematology results, the following order is suggested:

• HGB, HCT, WBC, BASO, EOS, LYM, MONO, NEUT, BASOLE, EOSLE, LYMLE, MONOLE, NEUTLE, RBC, PLAT.

Version: DRAFT ATH-1017-AD-0203 Confidential

### Table 14.3.4.3 Shift from Baseline to Post-Baseline Visits and Worst Post-Baseline Visit in Hematology Values Safety Population

#### Parameter: xxxx (units) (Low:<xxx/High:>xxx), (Low:<xxx/High:>xxx), (Low:<xxx/High:>xxx), (Low:<xxx/High:>xxx)

| | Worst Value During Study | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Baseline L | | Low Normal | | | Н | igh | Overall | |
| Treatment | Grade | n | (%) | n | (%) | n | (%) | n | (%) |
| Overall (N=xxx) | Low | xx | (xx.x) | XX | (xx.x) | ХХ | (xx.x) | xx | (xx.x) |
| overair (N-AAA) | Normal | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| | High | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| | Total | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |

- n: the number of participants who have values at both baseline (normal and abnormal) and post-baseline (abnormal).
- Baseline is defined as the last measurement prior to first dose.
- Overall column is the number of unique participants that have non-missing baseline values.
- Percentage for each grade is calculated using the number of participants in the Overall column.
- If a participant had a post-baseline value equal to LOW and another equal to HIGH, the participant is counted in each respective column.
- Low / Normal / High thresholds are based on the lower and upper limits of normal.
- Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y

#### Programming Notes:

- Replace highlighted Low/High with given low/high for parameter.
- For the subtitle of Parameter and the low/high values, if there are multiple reference ranges for a specific parameter, please display all range pairs.

#### NOTE:

- Worst value should be defined in the Protocol as low, high, or both or sponsor can confirm.
- If the missing category is not needed, then it can be omitted if a footnote is added specifying that only the participants with nonmissing baseline and at least 1 non-missing post-baseline are included. This table can be repeated for specific time points instead of "worst value during study".

Programming Notes:

- Please add missing rows or columns as per data requirements for completeness.
- The Visits will be displayed and also Worst Post-Baseline Visit <high/Low> assessment also displayed here.
- Please sort in this order: HGB, HCT, WBC, BASO, EOS, LYM, MONO, BASOLE, EOSLE, LYMLE, MONOLE, NEUTLE, RBC, PLAT.

Athira Pharma, Inc.

ATH-1017-AD-0203


Use the Table 14.3.4.3 shell.

NOTE: subset this table to show Chemistry lab parameters.

Programming Notes:

Table 14.3.4.9A

Shift from Baseline to Post-Baseline Visits in Urinalysis Values (Normal/Abnormal)

Safety Population

Use the Table 14.3.4.3 shell.

NOTE: subset this table to show Urinalysis lab parameters.

Table 14.3.4.9B

Shift from Baseline to Post-Baseline Visits and Worst Post-Baseline Visit in Urinalysis Values (Low/Normal/High)

Safety Population

Use the Table 14.3.4.3 shell.

NOTE: subset this table to show Urinalysis lab parameters.

Programming Notes:

Table 14.3.7.9

Summary of Liver Related Laboratory Abnormalities

Safety Population

| Parameter/Potentially<br>Clinically | 40 | mg ATH-1017<br>(N=xxx) | 70 | mg ATH-1017 | Overall (N=xxx) | |
|---|---|---|---|---|---|---|
| Significant Criterion | N1 | n (%) | N1 | n (%) | N1 | n (%) |
| Alanine Aminotransferase | XX | | XX | | XX | |
| <lln< td=""><td></td><td>xx (xx.x)</td><td></td><td>xx (xx.x)</td><td></td><td>xx (xx.x)</td></lln<> | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Normal (>=LLN - <=ULN) | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >1 - 3 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >3 - 5 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >5 - 10 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >10 - 20 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >20 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Aspartate Aminotransferase | XX | | xx | | xx | |
| <lln< td=""><td></td><td>xx (xx.x)</td><td></td><td>xx (xx.x)</td><td></td><td>xx (xx.x)</td></lln<> | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Normal (>=LLN - <=ULN) | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >1 - 3 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >3 - 5 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >5 - 10 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >10 - 20 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >20 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Alkaline Phosphatase | xx | | xx | | XX | |
| <lln< td=""><td>2121</td><td>xx (xx.x)</td><td>2121</td><td>xx (xx.x)</td><td>2121</td><td>xx (xx.x)</td></lln<> | 2121 | xx (xx.x) | 2121 | xx (xx.x) | 2121 | xx (xx.x) |
| Normal (>=LLN - <=ULN) | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >1 - 2 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >2 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Bilirubin | | | | | | |
| <t.t.n< td=""><td>XX</td><td>xx (xx.x)</td><td>XX</td><td>xx (xx.x)</td><td>XX</td><td>xx (xx.x)</td></t.t.n<> | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) |
| Normal (>=LLN - <=2 x ULN) | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| >2 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Hy's Law: ALT/AST>=3 x ULN and | | | | | | |
| BILI>=2xULN | XX | | XX | | XX | ( |
| Criteria Not Met | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| With ALP <2 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| With ALP >=2 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| ALP >=2 x ULN | XX | | XX | | XX | |
| Criteria Not Met | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| With ALT/AST <2 x ULN | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
With ALT/AST  $\geq$ 2 x ULN xx (xx.x) xx (xx.x) xx (xx.x)

- ULN: Upper Limit of Normal; LLN: Lower Limit of Normal. n = the number of participants with at least once post-baseline for the corresponding parameter. N1 = the number of participants who had at least 1 post-baseline assessment for the corresponding parameter; Percentages are based on N1. N: number of participants in the specified population for given treatment group.

- Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received. Participants with an abnormality in 70mg will be counted in the 70mg column. If that same participant switched to 40mg and reported an abnormality during the 40mg timeframe, that new abnormality is reported in the 40mg column. If the same abnormality reported while taking 40mg and 70mg then it is counted in both 40mg and 70mg groups; Overall is not a summation of the dose groups.

- Lab ranges between 201 and 203 differ due to differing lab vendors used.


Table 14.3.7.11
Summary of Eosinophil Lab Abnormalities
Safety Population

| Parameter | 40mg ATH-1017<br>(N=xxx) | 70mg ATH-1017<br>(N=xxx) | Overall (N=xxx) | |
|---|---|---|---|---|
| PCS Criterion | N1 n (%) | N1 n (%) | N1 | n (%) |
| Eosinophilia | xx | XX | xx | |
| Eosinophils >= 1500/uL | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Eosinophils >= 3000/uL | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Eosinophils >= 5000/uL | xx (xx.x) | xx (xx.x) | | xx (xx.x) |

<sup>-</sup> PCS: potentially clinically significant.

- n = the number of participants that met PCS criteria at least once post-baseline for the corresponding parameter.
- N1 = the number of participants who had at least 1 post-baseline assessment for the corresponding parameter; Percentages are based on N1.
- N: number of participants in the specified population for given treatment group.
- Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.
- Participants with an abnormality in 70mg will be counted in the 70mg column. If that same participant switched to 40mg and reported an abnormality during the 40mg timeframe, that new abnormality is reported in the 40mg column. If the same abnormality reported while taking 40mg and 70mg then it is counted in both 40mg and 70mg groups; Overall is not a summation of the dose groups.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


### Programming Notes:

• Split pages after 70mg group if doesn't fit

## **Vital Signs**

Version: DRAFT Confidential

Table 14.3.6.2
Potential Vital Signs Values of Concern at Any Time Post-Baseline Safety Population

| Vital Sign | 40 r | mg ATH-1017 | | ng ATH-1017 | | Overall |
|---|---|---|---|---|---|---|
| Abnormal Category | | (N=xxx) | | (N=xxx) | | (N=xxx) |
| | N1 | n (응) | N1 | n (응) | N1 | n (%) |
| Orthostatic Diastolic BP (mmHg) | XX | I | XX | l | XX | l |
| Standing Diastolic BP Decrease >=10mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Standing Diastolic BP Increase >=20mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Standing Diastolic BP >100mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Standing Diastolic BP >100 and Increase >=20mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Standing Diastolic BP <50 and Decrease >=10mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Standing Diastolic BP <50mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Orthostatic Systolic BP (mmHg) | xx | | XX | | XX | |
| Standing Systolic BP Decrease >=20mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Standing Systolic BP Increase >=20mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Standing Systolic BP >160mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Standing Systolic BP >160 and Increase >=20mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Systolic Blood Pressure (mmHg) | | | | | | |
| Systolic BP Decrease >=20mmHg | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) |
| Systolic BP Increase >=20mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Systolic BP >160mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Systolic BP >160 and Increase >=20mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Diastolic Blood Pressure (mmHg) | | | | | | |
| Diastolic BP Decrease >=10mmHg | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) |
| Diastolic BP Increase >=20mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Diastolic BP >100 and Increase >=20mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Diastolic BP <50 and Decrease >=10mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Diastolic BP >100mmHg | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Pulse Rate (beats/min) | xx | | XX | | XX | |
| Abnormal Heart Rate (<50 or >100 BPM) | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| Heart Rate Change >= 30 BPM | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |

- N1: the number of participants who have values at both baseline and post-baseline.
- Percentages are based on the Safety population. Participants may fall into more than one category.
- Participants with a potential value of concern in 70mg will be counted in the 70mg column. If that same participant switched to 40mg and reported a potential value of concern during the 40mg timeframe, that new potential value of concern is reported in the 40mg column. If the same potential value of concern reported while taking 40mg and 70mg then it is counted in both 40mg and 70mg groups; Overall is not a summation of the dose groups.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y

### Programming Notes:

• Visit can be added as a column to the left, if requested

## **ECG Tables**

# Table 14.3.7.4 ECG Interpretation at Any Time Post-Baseline Safety Population

| Parameter<br>Finding | 40 mg ATH-1017<br>(N=xxx)<br>n(%) | 70 mg ATH-1017<br>(N=xxx)<br>n(%) | Overall<br>(N=xxx)<br>n(%) |
|---|---|---|---|
| Interpretation - N1 | xxx | xxx | XXX |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- N1: the number of participants who have values at both baseline and post-baseline.
- N: number of participants in the specified population for given treatment group.
- Percentages are based on N1.
- A participant is counted only once for each finding category they fall into; if a participant has at least 1 abnormal record it is counted in the abnormal category.
- Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.
- Participants with an interpretation in 70mg will be counted in the 70mg column. If that same participant switched to 40mg and reported a interpretation during the 40mg timeframe, that new interpretation is reported in the 40mg column. If the same interpretation reported while taking 40mg and 70mg then it is counted in both 40mg and 70mg groups; Overall is not a summation of the dose groups.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


#### Programming Notes:

• Any abnormal finding for any post baseline visit will be counted as Abnormal.

Athira Pharma, Inc.

ATH-1017-AD-0203


# Table 14.3.7.5 Shift from Baseline to Post-Baseline Visits in ECG Values Safety Population

Use the Table 14.3.4.3 shell. NOTE: This table to show ECG parameters.

- Please add missing rows as per data requirements for completeness.
- Use "Visit (Timepoint)" concatenated in place of 'Visit" used in the Table 14.3.4.9A. The Visits will be displayed and also Worst Post-Baseline (Abnormal any time Post-Baseline) visitassessment also displayed here.

Version: DRAFT Confidential Table 14.3.7.6

## Table 14.3.7.6 Potential ECG Values of Concern at Any Time Post-Baseline Safety Population

| ECG Parameter Abnormal Category | | g ATH-1017<br>N=xxx) | 70 mg ATH-1017<br>(N=xxx) | | Overall (N=xxx) | |
|---|---|---|---|---|---|---|
| | N1 | n (%) | N1 | n (%) | N1 | n (%) |
| ECG Mean Heart Rate | XX | | XX | | XX | I |
| Heart Rate < 50 bpm | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| QRS Duration, Aggregate | XX | | XX | | XX | |
| QRS Duration > 120 msec | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| QRSAG Change > 25 msec | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| PR Interval, Aggregate | XX | | XX | | XX | |
| PR Interval > 250 msec | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| PRAG Change > 50 msec | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| QTcB Interval, Aggregate | XX | | xx | | xx | |
| QTcB Value >= 500 msec | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| QTcB Change >= 60 msec | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| QTcB Value >= 500 and Change >= 60 msec | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| QTcF Interval, Aggregate | XX | | xx | | XX | |
| QTcF Value >= 500 msec | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| QTcF Change >= 60 msec | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |
| QTcF Value >= 500 and Change >= 60 msec | | xx (xx.x) | | xx (xx.x) | | xx (xx.x) |

<sup>-</sup> ECG: Electrocardiogram; QRS: Quantronic Resonance System: PR: P-wave to QRS complex; QTcB: Heart rate-corrected QT Interval; QTcF: QT Interval Corrected using Fridericia's Formula; QRSAG: QRS Aggregate; N1: the number of participants who have values at both baseline and post-baseline.
- N: number of participants in the specified population for given treatment group. Percentages are based on N1. Participants may fall into more than one category. Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received. Participants with a potential value of concern in 70mg will be counted in the 70mg column. If that same participant switched to 40mg and reported a potential value of concern during the 40mg timeframe, that new potential value of concern is reported in the 40mg column. If the same potential value of concern reported while taking 40mg and 70mg then it is counted in both 40mg and 70mg groups; Overall is not a summation of the dose groups.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y

### **Concomitant Medications**

Table 14.3.8.2
Concomitant Medications by ATC Class and Preferred Name
Safety Population

| Anatomical Therapeutic Chemical Class (ATC)<br>Preferred Name | 40 mg ATH-1017<br>(N=xxx)<br>n(%) | 70 mg ATH-1017<br>(N=xxx)<br>n(%) | Overall<br>(N=xxx)<br>n(%) |
|---|---|---|---|
| Participants with at least 1 ATC class concomitant medication | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred name 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred name 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC Class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred name 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred name 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- ATC: Anatomical Therapeutic Chemical Class; WHO: World Health Organization. N: number of participants in the specified population for given treatment group. Percentages are based on N. A participant with multiple occurrences within an ATC class is counted only once. Concomitant medications (C) are defined as those medications used following the first administration of study drug. Medications started prior to the administration of study drug and continuing into the treatment period are considered as both prior and concomitant medications. WHO Drug Dictionary Version xx used for reporting of medications. Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received. Participants with a C in 70mg will be counted in the 70mg column. If that same participant switched to 40mg and reported a C during the 40mg timeframe, that new C is reported in the 40mg column. If the same C is reported while taking 40mg and 70mg then it is counted in both 40mg and 70mg groups; Overall is not a summation of the dose groups.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


### NOTE:

• Suggested sorting: ATC classes are presented alphabetically; PNs are sorted within ATC class in descending frequency in the Overall column.

#### Programming Notes:

• ATC2 and Preferred Term will be used for display.

## SECTION 16.X – PARTICIPANT DATA LISTINGS

## **Discontinued participants**

# Listing 16.2.1 Participant Disposition Safety Population

| Treatment | Participant<br>ID | AChEI<br>Usage/Age/<br>Sex/<br>Race | Site | First Dose Date | Last Dose Date (Day) | Date (Day) of<br>Completion or<br>Discontinuation | Completed or Primary Reason<br>Discontinued (Verbatim) |
|---|---|---|---|---|---|---|---|
| xxxxxxx | xxxxxxx | Y/xx/M/xx | XX | YYYY-MM-DD | YYYY-MM-DD (XX) | YYYY-MM-DD (XX) | Completed |
| xxxxxxx | xxxxxxx | N/xx/F/xx | XX | YYYY-MM-DD | YYYY-MM-DD (XX) | YYYY-MM-DD (XX) | Adverse event (Nausea) |
| xxxxxxx | xxxxxxx | N/xx/F/xx | XX | YYYY-MM-DD | YYYY-MM-DD (XX) | YYYY-MM-DD (XX) | Death |
| xxxxxxx | xxxxxxx | N/xx/F/xx | xx | YYYY-MM-DD | YYYY-MM-DD (XX) | YYYY-MM-DD (XX) | Other (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

<sup>-</sup> AChEI: Acetylcholinesterase inhibitor; M: Male; F: Female; Y: Yes; N: No;

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


- Please add time also if available.
- Treatment sorting order 40 mg ATH-1017, 70 mg ATH-1017

<sup>-</sup> Race Codes: 1: American Indian or Alaska Native; 2: Asian; 3: Black or African American; 4: Native Hawaiian or Other Pacific Islander; 5: White; 6: Other.

<sup>-</sup> Day is relative to the first dose date

<sup>-</sup> Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.

# Listing 16.2.1.1 Participants Reduced to 40mg Dose Safety Population

| Participant ID | AChEI<br>Usage/Age/<br>Sex/<br>Race | Parent Study<br>Treatment | Date of First<br>Dose | Date of Dose<br>Reduction (Day) | Reason for Dose<br>Reduction |
|---|---|---|---|---|---|
| xxxxxx | Y/xx/M/xx | ATH1017 xx<br>mg/Placebo | YYYY-MM-DD | YYYY-MM-DD (XX) | xxxxxxxx |
| XXXXXXX | N/xx/F/xx | ATH1017 xx<br>mg/Placebo | YYYY-MM-DD | YYYY-MM-DD (XX) | xxxxxxxxx |
| XXXXXXX | N/xx/F/xx | ATH1017 xx<br>mg/Placebo | YYYY-MM-DD | YYYY-MM-DD (XX) | xxxxxxxxx |
| xxxxxxx | N/xx/F/xx | ATH1017 xx mg/Placebo | YYYY-MM-DD | YYYY-MM-DD (XX) | xxxxxxxx |

<sup>-</sup> Day is relative to first dose date.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


- Only include participants with ADSL.DOSE40MG='Y'
- Please add time also if available.

<sup>-</sup> M: Male; F: Female; Y: Yes; N: No; AChEI: Acetylcholinesterase inhibitor

<sup>-</sup> Source of dose reduction data to be added as footnote

<sup>-</sup> Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.

## **Protocol deviations**

# Listing 16.2.2 Major Protocol Deviations Safety Population

| | Participant | AChEI<br>Usage/Age/<br>Sex/ | Date of Deviation | | |
|---|---|---|---|---|---|
| Treatment | ID | Race | (Day) | Category | Descriptions |
| xxxxxxx | xxxxxxx | Y/45/M/xxxx | YYYY-MM-DD (XX) | xxxxxxxxxx | xxxxxxxxxxxxxxxxxxx |
| | | | YYYY-MM-DD (XX) | XXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | YYYY-MM-DD (XX) | XXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXX |
| xxxxxxx | xxxxxxx | N/49/F/xxxx | YYYY-MM-DD (XX) | xxxxxxxxx | xxxxxxxxxxxxxxxxx |

<sup>-</sup> AChEI: Acetylcholinesterase inhibitor; M: Male; F: Female; Y: Yes; N: No;

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


- Please add time also if available.
- Only Major deviations will be displayed.
- Treatment sorting order 40 mg ATH-1017, 70 mg ATH-1017

<sup>-</sup> Race Codes: 1: American Indian or Alaska Native; 2: Asian; 3: Black or African American; 4: Native Hawaiian or Other Pacific Islander; 5: White; 6: Other.

<sup>-</sup> Day is relative to the first dose date.

<sup>-</sup> Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.

**Demographics and Baseline Characteristics** 

Listing 16.2.4.1
Participant Demographics and Baseline Characteristics
Safety Population

| Treatment | Participant<br>ID | AChEI<br>Usage/Age/<br>Sex/Race | Ethnicity | Weight<br>(kg) | Height<br>(cm) | BMI<br>(kg/m2) | Years of<br>Education |
|---|---|---|---|---|---|---|---|
| xxxxxxx | xxxxxxx | Y/xx/M/xx | Not Hispanic<br>or Latino | XX | XX | XX | xx |
| xxxxxxx | xxxxxxx | N/xx/F/xx | Not Hispanic<br>or Latino | XX | XX | XX | xx |

<sup>-</sup> BMI: Body Mass Index; AChEI: Acetylcholinesterase inhibitor; M: Male; F: Female; Y: Yes; N: No;

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


Programming Notes:

.

<sup>-</sup> Race Codes: 1: American Indian or Alaska Native; 2: Asian; 3: Black or African American; 4: Native Hawaiian or Other Pacific Islander; 5: White; 6: Other.

<sup>-</sup> Baseline is defined as the last measurement prior to first dose for safety endpoints, and either the measurement on Day 1, or else the last measurement before Day 1 if there is no Day 1 measurement for efficacy endpoints.

<sup>-</sup> Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.

# Listing 16.2.6 Prior and Concomitant Medications Safety Population

| Treatment | Participant<br>ID | P/C | ATC Level 3/<br>Preferred name/<br>Reported name | Start Date/Time<br>(Day)/<br>End Date/Time (Day) /<br>Ongoing | Indication | Dose and units | Frequency | Route |
|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xxxxxxx | Х | xxxxxx/<br>xxxxxxxxxxx/<br>xxxxxxxxxxxxx | YYYY-MM-DD HH:MM (XX)/ YYYY-MM-DD HH:MM (XX) | HYPERTENSION | xxx mg | QD | ORAL |
| xxxxxxx | xxxxxxx | X | ************************************** | YYYY-MM-DD HH:MM (XX) (XX)/ YYYY-MM-DD HH:MM (XX) | DIABETES | xxx mg | QD | ORAL |

- P: Prior Medication; C: Concomitant Medication; ATC: Anatomical Therapeutic Chemical.
- Day is relative to the first dose date.
- Prior medications (P) are defined as those medications used prior to the administration of study drug.
- Concomitant medications (C) are defined as those medications used following the first administration of study drug. Medications started prior to the administration of study drug and continuing into the treatment period are considered as both prior and concomitant medications.
- WHO Drug Version xx.x was used for reporting of prior and concomitant medications.
- Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.
- '/' for End Date (Day) means no date was provided.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


Programming Notes:

•

## LAB/ECG/VS LISTINGS

Listing 16.2.8.1
Chemistry Laboratory Values Where at Least One Value is a Potential Value of Concern

Safety Population

| | | | | | Phosp | aline<br>hatase<br>/L) | Aminotr | anine<br>ansferase<br>J/L) | Aminotra | rtate<br>insferase<br>/L) | | rubin<br>ol/L) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Participant<br>ID | AChEI<br>Usage/<br>Age/Sex/<br>Race | Study<br>Visit | Collection<br>Date/Time (Day) | Observed<br>Value | Change<br>from<br>Baseline | Observed<br>Value | Change<br>from<br>Baseline | Observed<br>Value | Change<br>from<br>Baseline | Observed<br>Value | Change<br>from<br>Baseline |
| XXX xxx | xxxxxx | Y/xx/M/xx | xxxx | YYYY-MM-<br>DDTHH:MM (XX) | xx.xx* | xx.xx | xx.x* | XX.X | xx.xxx* | xx.xxx | xx.xxx* | xx.xx |
| | | | xxxx | YYYY-MM-<br>DDTHH:MM (XX) | XX.XX | XX.XX | XX.X | XX.X | xx.xxx | xx.xxx | XX.XXX | xx.xxx |
| | | N/xx/F/xx | XXXX | YYYY-MM-<br>DDTHH:MM (XX) | XX.XX | XX.XX | XX.X | XX.X | XX.XXX | XX.XXX | XX.XXX | XX.XXX |

<sup>-</sup> AChEI: Acetylcholinesterase inhibitor; Y: Yes; N: No; M: Male; F: Female;

- Baseline is defined as the last measurement prior to first dose.
- Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


- Use code for race.
- Where at least one value for that patient is marked as high or low. Display baseline only if there are High or Low values.
- Run for all Chemistry variables (Albumin (g/L), Alkaline Phosphatase (U/L), Aspartate Aminotransferase (U/L), Bilirubin (umol/L), Calcium (mmol/L), Chloride (mmol/L), Cholesterol (mmol/L), Creatine Kinase (U/L), Creatinine (umol/L), Gamma Glutamyl Transferase (U/L), Glucose (mmol/L), HDL Cholesterol (mmol/L), Hemoglobin AlC (%), LDL Cholesterol (mmol/L), Potassium (mmol/L), Protein (g/L), Protein (g/L), Sodium (mmol/L), Triglycerides (mmol/L).

<sup>-</sup> Race Codes: 1: American Indian or Alaska Native; 2: Asian; 3: Black or African American; 4: Native Hawaiian or Other Pacific Islander; 5: White; 6: Other.

<sup>- \*</sup>Indicates Baseline.

# Listing 16.2.8.2 Hematology Laboratory Values Where at Least One Value is a Potential Value of Concern Safety Population

- Repeat Listing 16.2.8.1 where at least one value for that patient is marked as high or low.
- Run for all Hematology variables (Basophils (10^9/L), Basophils/Leukocytes (fraction of 1), Eosinophils (10^9/L), Eosinophils/Leukocytes (fraction of 1), Erythrocytes (10^12/L), Hematocrit (fraction of 1), Hemoglobin (g/L), Leukocytes (10^9/L), Lymphocytes (10^9/L), Lymphocytes (10^9/L), Lymphocytes/Leukocytes (fraction of 1), Monocytes (10^9/L), Monocytes/Leukocytes (fraction of 1), Platelets (10^9/L)).

# Listing 16.2.8.3 Vital Signs Values Where at Least One Value is a Potential Value of Concern Safety Population

 Repeat Listing 16.2.8.1 where at least one value for that patient is marked as high or low. To identify potential value of concerns, please use the criteria shown below:

```
Orthostatic Diastolic BP (mmHq)
  Standing Diastolic BP Decrease >=10mmHg
  Standing Diastolic BP Increase >=20mmHg
  Standing Diastolic BP >100mmHg
  Standing Diastolic BP >100 and Increase >=20mmHg
  Standing Diastolic BP <50 and Decrease >=10mmHg
  Standing Diastolic BP <50mmHg
Orthostatic Systolic BP (mmHg)
  Standing Systolic BP Decrease >=20mmHg
  Standing Systolic BP Increase >=20mmHg
  Standing Systolic BP >160mmHg
  Standing Systolic BP >160 and Increase >=20mmHg
Systolic Blood Pressure (mmHq)
  Systolic BP Decrease >=20mmHg
  Systolic BP Increase >=20mmHg
  Systolic BP >160mmHg
  Systolic BP >160 and Increase >=20mmHg
Diastolic Blood Pressure (mmHg)
  Diastolic BP Decrease >=10mmHg
  Diastolic BP Increase >= 20mmHg
  Diastolic BP >100 and Increase >=20mmHg
  Diastolic BP <50 and Decrease >=10mmHg
```

Diastolic BP >100mmHg Diastolic BP <50mmHg

Pulse Rate (beats/min)
 Abnormal Heart Rate (<50 or >100 BPM)
 Heart Rate Change >= 30 BPM

 $\qquad \qquad \text{ Listing 16.2.9}$  ECG Parameters Where at Least One Value is a Potential Value of Concern

Safety Population

| Treatment | Participant<br>ID | AChEI Usage/<br>Age/Sex/<br>Race | Study Visit | Collection Date/Time (Day) | Parameter (unit) | Abnormality |
|---|---|---|---|---|---|---|
| XXX | xxxxxxx | Y/xx/M/xx | xxxx | YYYY-MM-DDTHH:MM (XX)* | xx (xx) | xxxxxxxx |
| | AAAAAA | 1/ XX/ 11/ XX | AAAA | IIII PHA DDIIII.PHA (MM) | xx (xx) | XXXXXXXX |
| | | | | xx (xx) | mmmmm | |
| | | | | | xx (xx) | |
| | | | | | xx (xx) | |
| | | | | | xx (xx) | |
| | | | | | xx (xx) | xxxxxxxx |
| | | | | | xx (xx) | xxxxxxxx |
| | | | xxxx | YYYY-MM-DDTHH:MM (XX) | xx (xx) | xxxxxxxx |
| | | | | | xx (xx) | xxxxxxxx |
| | | | | | xx (xx) | XXXXXXXX |
| | | | | | xx (xx) | |
| | | | | | xx (xx) | |
| | | | | | xx (xx) | XXXXXXXX |
| | | | | | xx (xx) | XXXXXXXX |
| | | | | | xx (xx) | |
| | | | | | xx (xx) | XXXXXXXX |

<sup>-</sup> ECG: Electrocardiogram.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y


### Programming Notes:

• If at least one parameter has an abnormality for that visit, print all non-missing parameters for that visit, filling in the abnormality column when applicable. Display baseline only if there are abnormal findings.

<sup>- \*</sup>Indicates Baseline.

<sup>-</sup> Baseline is defined as the last measurement prior to first dose.

## STANDARD FIGURE SHELLS

Figure 14.3-1.1
eDISH (evaluation of Drug Induced Serious Hepatotoxicity)
Safety Population



<sup>-</sup> ALT = Alanine Aminotransferase; AST = Aspartate Aminotransferase; ULN = upper limit of normal. All values were normalized to the ULN that was provided for each participant, lab parameter, and visit. Data displayed in this figure represents the original result as a proportion of ULN.

Generated from program.sas on DDMMMYYYY HH:MM:SS. Source dataset(s): ADxx. Date of data extraction: DDMMMYYYY.

Page X of Y

#### Programming Notes:

• 40mg Ath-1017 and 70mg Ath-1017 (no Placebo due to Placebo not in study).

<sup>-</sup> Values are the maximum post-baseline. ALT/AST is the maximum Upper Limit of Normal of either ALT or AST.

<sup>-</sup> Participants with a value in 70mg will be counted in the 70mg group. If that same participant switched to 40mg and reported a value during the 40mg timeframe, that new value is reported in the 40mg group. If the same value is reported while taking 40mg and 70mg then it is counted in both 40mg and 70mg groups; Safety population includes all participants who received at least one dose of study medication, classified by actual treatment received.